CLINICAL TRIAL: NCT07228546
Title: The Effects of Demographic and Clinical Data of Patients on the Assessment of Cerebral Oxygen Monitoring Values Applied During Coronary Artery Bypass Grafting
Brief Title: The Effects of Demographic and Clinical Data of Patients on Cerebral Oxygen Monitoring Values
Status: Completed | Type: Observational
Sponsor: Tuna Şahin (Other)
Responsible Party: Sponsor-Investigator, Tuna Şahin, Anesthesiologist, Adana City Training and Research Hospital
Organization: Adana City Training and Research Hospital (Other)
Other Study IDs: Adana City TRH
Record Dates: First submitted 2025-09-30; First posted 2025-11-14 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Oxygen Saturation
Keywords: near infrared spectroscopy; coronary artery bypass grafting; regional cerebral oxygen saturation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to examine the effects of patients' clinical and demographic datas on cerebral oxygen saturation values. Brain oxygenation is measured using near infrared spectroscopy (NIRS). The primary outcome measure of the study is the regional oxygen saturation (rSO2) values measured on the monitor at twelve time points. The other primary outcome measures consist of baseline arterial and venous blood gas analysis and baseline activated clotting time measurements.

DETAILED DESCRIPTION:
This prospective observational study analyzes 80 patients between the ages of 25-80 years who are undergoing elective coronary artery bypass grafting (CABG) surgery. Demographic data of the patients such as age, gender, comorbidities, body mass index are recorded. In addition to standard monitoring, cerebral oximetry monitoring (NIRS) is applied to the patients. Baseline arterial and venous blood gas analysis values, baseline activated clotting time measurements are recorded. Durations of anesthesia, surgery , cardiopulmonary bypass , aortic cross- clamping are recorded. Time points for rSO2 values are baseline, induction, sternotomy, cannulation, pump entry, cross clamp placement, 34º C ,36º C, lowest temperature, cross clamp removal, pump exit, skin closure.

ELIGIBILITY:
Inclusion criteria:

* Accepting to participate in the study
* Undergoing elective coronary artery bypass grafting surgery
* Age 25-80 years Ejection fraction 30% and above

Exclusion criteria:

* Non volunteers
* Age <25 or >80 years
* Ejection fraction below 30%
* Patients with history of neurological disease or neurosurgery
* Emergency surgery
* Concurrent valve surgery
* Patients with history of carotid artery stenosis
* Patients with need for preoperative intraaortic balloon pump or inotropic support

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective coronary artery bypass grafting surgery
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2025-05-12 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Regional oxygen saturation values | Baseline and peroperative measurements until the and of surgery
  Regional oxygen saturation values measurement at twelve points.
Baseline arterial blood gas analysis | Within 5 minutes after arterial cannulation for the baseline measurement
  The baseline arterial blood gas sample taken from the patient after arterial cannulation
Venous blood gas analysis | Within 5 minutes after central jugular venous cannulation
  Venous blood gas sample taken from the patient after central jugular venous cannulation
Baseline activated clotting time measurement | Within 5 minutes after arterial cannulation for the baseline measurement
  The baseline measurement of activated clotting time after arterial cannulation

CONTACTS AND LOCATIONS:
Locations (1):
- Tuna Şahin, Adana, Yüreğir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No